CLINICAL TRIAL: NCT01953159
Title: Validation of a Polygenic Neurotoxicity Risk Score in Patients With Unusually Severe Paclitaxel-Induced Neuropathy
Brief Title: Assessment of Paclitaxel-Induced Neuropathy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB13-0775
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood, DNA,Peripheral Blood Mononuclear Cells (PBMC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with severe neuropathy: Patients with severe neuropathy after treatment with paclitaxel. Blood samples and patient questionnaires will be collected.
  Interventions: Other: Blood Collection; Other: Patient Questionnaires
- Patients without neuropathy: Patients will be enrolled to this cohort and matched to a specified subject with neurotoxicity based on age (within 10 years), tumor type, chemotherapy regimen or total paclitaxel dosage, race, and ethnicity
  Interventions: Other: Blood Collection; Other: Patient Questionnaires

INTERVENTIONS:
Other: Blood Collection
Other: Patient Questionnaires

SUMMARY:
The purpose of this study is to collect clinical data, blood samples, and self reported symptoms from patients that experience unusually severe neuropathy after treatment with paclitaxel. This data will be used to develop predictive markers for neuropathy. Blood samples will be used to create induced pluripotent stem (iPS) cells and eventually artificial nerve cells to be used to study neuropathy in the lab.

ELIGIBILITY:
Inclusion Criteria (Severe Toxicity Group):

* Diagnosis of cancer (including, but not limited to, breast and ovarian cancer)
* Females aged 18 and older
* History of grade 3 or higher peripheral neurotoxicity, any neuromotor, neurocortical, or neurocerebellar toxicity, myalgias or arthralgias refractory to non-steroidal anti-inflammatory drugs and steroids, ong-term persistence (> 6 months) of grade 2 or higher peripheral neuropathy, or other unusually severe neurotoxicity approved for inclusion in study by Principal Investigator after completion of paclitaxel chemotherapy regimen or history of peripheral neuropathy that required treatment with narcotics or grade 2 or higher peripheral neuropathy after only 1 to 2 doses of paclitaxel.

Inclusion Criteria (Control Group):

* History of no neurotoxicity (grade 0) after completion of a standard paclitaxel-containing chemotherapy regimen
* Females age 18 and older
* Matched to a specified subject with neurotoxicity based on age (within 10 years), tumor type, chemotherapy regimen or total paclitaxel dosage, race, and ethnicity

Exclusion Criteria :

* Treatment with other severely neurotoxic chemotherapy (i.e. cisplatin) prior to or concomitantly with paclitaxel. Carboplatin therapy is allowed.
* Presence of peripheral neuropathy prior to paclitaxel therapy
* Poorly controlled or insulin-dependent diabetes or other condition likely to predispose to neurotoxicity (alcoholism, Charcot-Marie-Tooth disease)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated with paclitaxel
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-08-29 (Actual); Primary Completion 2027-05-19 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Validation of polygenic risk score | 2 years
  Patients will be assessed for neuropathy symptoms and blood samples will be analyzed to detect potential predictive markers

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States